CLINICAL TRIAL: NCT06301659
Title: Impact of Adapted Mirror Therapy on Individuals With Hemiparesis of the Upper Limb Following a Stroke: A Randomized Controlled Trial
Brief Title: Impact of Adapted Mirror Therapy on Individuals With Hemiparesis of the Upper Limb Following a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmadu Bello University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Jingxiang-Jiu
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified mirror therapy+routine rehabilitation therapy (Experimental): The study lasted 30 days for each participant. The patients enrolled were randomly divided into the experimental group and the control group, all under routine rehabilitation therapy. Additionally, the patients in the experimental group were given modified mirror therapy.
  Interventions: Behavioral: routine rehabilitation therapy; Behavioral: Modified mirror therapy
- routine rehabilitation therapy (Active Comparator): The study lasted 30 days for each participant. The patients enrolled were randomly divided into the experimental group and the control group, all under routine rehabilitation therapy.
  Interventions: Behavioral: routine rehabilitation therapy

INTERVENTIONS:
Behavioral: routine rehabilitation therapy — The Participants with stable vital signs were scheduled for specialized rehabilitation training upon enrollment, and targeted rehabilitation programs were selected based on the patient's specific limb function impairment, conducted by experienced rehabilitation therapists.
Behavioral: Modified mirror therapy — The patients were instructed to watch the recorded video and imitate the movements of their affected limbs. After the video ended, only the instructions and synchronized music were played. The patient was required to sit in front of a mirror table, with the mirror placed between both arms and facing the healthy side. The patient was required to recall the video based on the verbal instructions while using the healthy side to perform movement training. They were also asked to observe the reflected motion of the healthy limb in the mirror, simultaneously imagining the affected limb moving in sync (the patient focused on the front of the mirror, avoiding direct eye contact with the healthy hand, to create the sensation that it was the affected hand performing the movements).
  Arms: modified mirror therapy+routine rehabilitation therapy

SUMMARY:
Patients with upper limb hemiplegia after stroke, who were admitted in the Department of Rehabilitation Medicine, were enrolled. The study lasted 30 days for each participant. The patients enrolled were randomly divided into the experimental group and the control group, all under routine rehabilitation therapy. Additionally, the patients in the experimental group were given modified mirror therapy. On day 1 and day 30, patients' Upper Limb function were compared.

DETAILED DESCRIPTION:
Upper limb hemiparesis is a motor and sensory disorder that occurs after stroke, with an incidence rate of up to 55% to 75%. This was a Randomized controlled trial. Patients with upper limb hemiplegia after stroke, who were admitted in the Department of Rehabilitation Medicine, were enrolled. The study lasted 30 days for each participant. The patients enrolled were randomly divided into the experimental group and the control group, all under routine rehabilitation therapy. Additionally, the patients in the experimental group were given modified mirror therapy. On day 1 and day 30, patients' Upper Limb function were compared.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of stroke.
* The first-onset stroke.
* Presenting with unilateral upper limb dysfunction, within Brunnstrom stage Ⅱ to Ⅳ on the affected side, and Ash-worth score ≤2.
* No obvious cognitive impairment, with Mini-Mental State Examination (MMSE) score >21 points.
* National Institutes of Health Stroke Scale (NIHSS) score >4 points.
* Stable vital signs, no severe diseases such as cancer, liver or kidney disorders.
* Aged 35-70 years.
* Courses of diseases 2-6 weeks.

Exclusion Criteria:

* Presence of aphasia, apraxia, or hemispatial neglect.
* Presence of hearing, vision, or comprehension impairments that hinder diagnosis and treatment.
* Complicate with traumas, fractures, or other progressive neuro-muscular system diseases.
* Severe spasticity in the upper limbs.
* Severe bone, joint, or muscle deformities or lesions.
* History of mental illness.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity | day 1 and day 30
  The Fugl-Meyer Assessment-Upper Extremity was used to evaluate the patient's upper limb function and motor control. It included the assessment of movements in the shoulder, elbow joint, wrist, and fingers. During the assessment, the assessor observed and recorded the patient's abilities and limitations in specific actions. Based on the patient's performance in each sub-item, the assessor assigned a score using a 0-2 scale, a score of 0 indicating inability to perform, 1 indicating partial ability, and 2 indicating full ability. Finally, the scores for each sub-item were summed up to obtain an overall upper limb function score of 0-66, with scores positively correlated with the upper limb function.

SECONDARY OUTCOMES:
coordinated contraction rate-Surface electromyography | day 1 and day 30
  The surface electromyography (sEMG) was used to assess the coordinated contraction rates of the biceps brachii on the affected upper limb. The surface electromyography device was used for detection, with the most prominent part of muscle belly of the biceps brachii serving as the monitoring points. During the maximum isometric voluntary contraction (MIVC) state of elbow flexion or extension, two channels were used to separately record the integrated electromyographic values (iEMG) of the biceps brachii, and the antagonists. Measurements were taken three times to obtain the maximum value, and the coordinated contraction rate (CR) during elbow flexion or extension under MIVC conditions was calculated using the formula: CR (%) = Antagonist muscle iEMG / (Agonist muscle iEMG + Antagonist muscle iEMG).
Visual Analog Scale | day 1 and day 30
  the pain level of the affected shoulder was measured using the Visual Analog Scale (VAS), with 0 indicating no pain and 10 indicating unbearable severe pain. The lower score indicated the lighter pain.
Anxiety | day 1 and day 30
  The anxiety was assessed using the Generalized Anxiety Disorder-7 (GAD-7), including items related to fear, worry, attention, etc. The total score ranged from 0 to 21, which was positively correlated with potential anxiety. In the previous study, the GAD-7 scale demonstrated a Cronbach's α-coefficient of 0.879. The scores range from 0 to 21. The higher scores mean a worse outcome.
Depression | day 1 and day 30
  The depression was assessed using the Patient Health Questionnaire-9 (PHQ-9), with aspects including mood swings, optimism, sleep quality, appetite, etc. The total score of PHQ-9 ranged from 0 to 27, which was positively correlated with potential depression. In the previous study, the PHQ-9 scale demonstrated a Cronbach's α-coefficient of 0.913.The scores range from 0 to 27.The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group
Locations (1):
- Affiated Hos., Huabei, China